CLINICAL TRIAL: NCT05688748
Title: Effectiveness Evaluation of a Dengue Self-monitoring System (DeSMoS) to Reduce Treatment Delay in Malaysia
Brief Title: Effectiveness Evaluation of a Dengue Self-monitoring System
Acronym: DeSMoS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022328-11112
Record Dates: First submitted 2023-01-05; First posted 2023-01-18 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Dengue
Keywords: dengue; outpatient care; self-monitoring system; treatment delay; warning symptoms
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dengue monitoring system (Experimental): The participants will be given access to download a dengue self-monitoring application and use the application at home to key in their symptoms, three times a day throughout their outpatient follow up for dengue.
  Interventions: Other: Dengue self-monitoring system
- Usual care (No Intervention): Patients will be managed as per usual outpatient care for dengue in the clinic.

INTERVENTIONS:
Other: Dengue self-monitoring system — The system has a symptom monitoring algorithm whereby patient would be asked to report their symptoms thrice daily (9am, 2pm and 8pm). The algorithm is developed by the researchers which consist of primary care doctors, emergency physician and infectious disease specialists. If the patient reports warning symptoms (persistent vomiting, persistent diarrhoea, abdominal pain, bleeding, difficulty breathing, feel like fainting, difficulty carrying out usual activities, drowsiness, reduced urine output and reduced urine output), the system will advise patients to seek earlier medical care instead of waiting for the scheduled appointment the next day/other days.
  Other Names: DeSMoS
  Arms: Dengue monitoring system

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of a dengue self-monitoring system with standard care in reducing treatment delay among dengue patients receiving outpatient care. The main question it aims to answer are:

• Is a dengue self-monitoring system effective in reducing treatment delay in dengue patients? Participants will use the dengue monitoring system in addition to the standard care they are receiving for outpatient follow up for dengue.

Researchers will compare them with dengue patients receiving the usual standard care to see if the dengue monitoring system reduces delay in treatment seeking in patients.

DETAILED DESCRIPTION:
Dengue Self-Monitoring System (DeSMoS) was developed to guide patients about warning signs and advise them to visit a doctor appropriately before their scheduled follow up on the next day, apart from motivating them to comply to the daily follow up visits at the clinic. DeSMoS is hypothesised to effectively reduce delay in treatment seeking in dengue patients.

The main aim of this system is to get dengue patients to key-in their symptoms regularly via the app when they are at home. Reminders will appear on the phone to remind them to key in the symptoms thrice daily.

The system is designed as a supportive tool for outpatient dengue management. It is not meant to replace to usual standard care for dengue care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old and above
* Newly diagnosed with dengue fever
* Have a smartphone
* Receiving outpatient follow up for dengue

Exclusion Criteria:

* Hearing and speech impairment
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Reduction in treatment delay | Up to two weeks
  Proportion of patients with warning symptoms who return to see a doctor earlier than scheduled

SECONDARY OUTCOMES:
Compliance to follow up | Up to two weeks
  Proportion of patients who are compliant of all follow up visits
Development of warning symptoms | Up to two weeks
  Proportion of patients who develop warning symptoms
Hospitalization | Up to two weeks
  Proportion of patients with warning symptoms who are admitted to hospital

CONTACTS AND LOCATIONS:
Overall Officials: Wei Leik Ng, Principal Investigator — University of Malaya
Locations (1):
- Klinik Kesihatan Seksyen 7 Shah Alam, Shah Alam, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Leo YS, Gan VC, Ng EL, Hao Y, Ng LC, Pok KY, Dimatatac F, Go CJ, Lye DC. Utility of warning signs in guiding admission and predicting severe disease in adult dengue. BMC Infect Dis. 2013 Oct 24;13:498. doi: 10.1186/1471-2334-13-498. PMID 24152678
- [Result] Herbuela VRDM, Karita T, Francisco ME, Watanabe K. An Integrated mHealth App for Dengue Reporting and Mapping, Health Communication, and Behavior Modification: Development and Assessment of Mozzify. JMIR Form Res. 2020 Jan 8;4(1):e16424. doi: 10.2196/16424. PMID 31913128